CLINICAL TRIAL: NCT03856879
Title: AdvanCing High-quality COPD Care for People With Immune Dysfunction by Implementing EVidence-based Management Through Proactive E-consults
Brief Title: High-quality COPD Care for People With Immune Dysfunction Through Proactive E-consults
Acronym: ACHIEVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: VA Puget Sound Health Care System (U.S. Federal Agency); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); VA Eastern Colorado Health Care System (U.S. Federal Agency); University of Colorado, Denver (Other); VA Greater Los Angeles Healthcare System (U.S. Federal Agency); Atlanta VA Medical Center (U.S. Federal Agency); Yale University (Other); VA Connecticut Healthcare System (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); VA Tennessee Valley Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1U01HL142103-01 (NIH)
Record Dates: First submitted 2019-02-20; First posted 2019-02-27 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: COPD; HIV/AIDS
Keywords: Chronic obstructive pulmonary disease; intervention studies; randomized controlled trial; provider satisfaction; patient satisfaction; E-consult
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Acquired Immunodeficiency Syndrome; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Providers will be randomly assigned to the intervention or control group, stratified by site, provider type and panel size.
Who Masked: Outcomes Assessor
Masking Description: Study staff conducting patient surveys and evaluating quality of COPD care will be blinded to intervention/control assignment of the patient's provider.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual care (No Intervention): Providers in this arm will provide usual care to their HIV+ patients with COPD.
- Proactive E-consult (Experimental): Providers in this arm will receive proactive E-consults with expert recommendations for COPD care prior to appointments with HIV+ patients with COPD.
  Interventions: Behavioral: Proactive E-consult

INTERVENTIONS:
Behavioral: Proactive E-consult — E-consult recommendations and orders will be developed by a panel of pulmonologists and will address a range of care elements for patients with COPD.
  Arms: Proactive E-consult

SUMMARY:
This study examines an intervention to promote effective, evidence-based care and de-implement inappropriate therapies for COPD in HIV-infected (HIV+) patients. The intervention facilitates specialist support of primary care, which includes infectious disease (ID) physicians who serve as the primary care providers (PCP) for their HIV+ patients in the ID clinic. Rather than relying on referral-driven specialty care which may be a barrier to access, pulmonologists will proactively support ID providers to manage a population of HIV+ patients with COPD, delivering real-time evidence-based recommendations tailored to the individual HIV+ patient in the form of an E-consult.

DETAILED DESCRIPTION:
Emerging data support that barriers to high quality COPD care are likely accentuated in HIV+ persons. Taken together, decreased recognition of smoking, lack of referral for pulmonary evaluation, worse symptoms and greater exacerbation rates point towards low quality of care for COPD in HIV+ patients. Our preliminary data supports that COPD is inadequately managed in HIV+ patients. These data demonstrate that current management of COPD in HIV+ patients do not adhere to guidelines, that ICS may be over-prescribed and long-acting bronchodilators under-utilized, and support the need to improve evidence-based COPD care in HIV+ patients. Appropriate use of COPD therapies is particularly important for HIV+ patients, as side effects and toxicities could be more harmful in HIV+ patients, given their concomitant multimorbidity and polypharmacy. In summary, an intervention to improve the evidence-based delivery of COPD care can improve outcomes for HIV+ patients. Benefits may extend beyond COPD-related measures. Appropriate use of COPD controller medications can decrease symptoms and exacerbations, and improve health-related quality of life. Our proposed study to has a high potential to substantially improve the quality of care for COPD and patient-centered outcomes for a large number of HIV+ Veterans.

This study tests an intervention to promote effective, evidence-based care and de-implement inappropriate therapies for COPD in HIV+ patients. The intervention facilitates specialist support of primary care, which includes infectious disease (ID) physicians who serve as the primary care providers (PCP) for their HIV+ patients in the ID clinic. Rather than relying on referral-driven specialty care, which may be a barrier to access, pulmonologists will proactively support ID providers to manage a population of HIV+ patients with COPD, delivering real-time evidence-based recommendations tailored to the individual HIV+ patient. The investigators will leverage the Department of Veterans Affairs (VA) clinical and informatics infrastructures to communicate between intervention-team members developing the recommendations (using VA Extension for Community Health Outcomes [ECHO]) and to patients' clinical providers through the electronic health record (EHR) as an E-consult. To limit the burden on the provider, the intervention team will draft recommendations as preliminary orders for providers to review. To preserve their autonomy, the provider has the discretion to endorse (sign), modify or cancel the orders.

This study uses a two-arm cluster randomized controlled trial intervention design grounded in the chronic care model with outcomes evaluated using the RE-AIM (Reach, Effectiveness, Adoption, Implementation and Maintenance) framework. The investigators will evaluate barriers and facilitators of optimal COPD care for HIV+ patients, and of effective adoption, implementation and maintenance of the proactive E-consult program, guided by the Consolidated Framework for Implementation Research (CFIR).

This study involves the recruitment and enrollment of two populations: providers and patients. Providers will be recruited at the beginning of the study; providers that enroll will be randomly chosen to either provide usual care (control) or to receive E-consults for their HIV+ patients with COPD (intervention). Patients of enrolled providers will be recruited after attending an appointment with their provider. Enrolled patients will be asked to complete a set of surveys, and some patients will be offered the opportunity to participate in an interview about their care.

ELIGIBILITY:
Inclusion criteria:

Providers:

• Outpatient infectious disease providers at one of the seven local sites participating in this study.

Patients:

• HIV+ patients with COPD treated by providers enrolled in the study.

Exclusion Criteria:

Providers:

• Trainees

Patients:

• Significant cognitive dysfunction, language barriers or severe psychiatric disorder, impairing ability to participate in surveys and interviews.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
% of COPD care recommendations received by patients of enrolled providers | 6 months following provider/patient appointment
  % of COPD care recommendations received by the patient, examined collectively for each patient and individually by type of recommendation (e.g. use of spirometry, long acting bronchodilator, smoking cessation, vaccination, etc.) to assess the overall quality of COPD care.

SECONDARY OUTCOMES:
Patient health-related quality of life | 6 weeks following provider/patient appointment
  Patient-reported health-related quality of life on the Medical Outcomes 12-item short form (SF-12), a patient self-report survey. This survey is a 12-item scale with two subscales (mental and physical components). Summary scores range from 0-100, with higher scores reflecting better health.

OTHER OUTCOMES:
HIV provider satisfaction with specialty-care support | Baseline: prior to intervention roll-out. Follow-up: after exposure to intervention (defined as having received at least 2 E-consults), up to 3 years.
  Baseline and follow-up self-report surveys (all participating providers) and interviews (sample of providers)

CONTACTS AND LOCATIONS:
Overall Officials: David H. Au, MD, MS, Principal Investigator — VA Puget Sound Health Care System; Kristina A. Crothers, MD, Principal Investigator — VA Puget Sound Health Care System; Christian D. Helfrich, PhD, MPH, Principal Investigator — VA Puget Sound Health Care System
Locations (7):
- United States (7):
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - VA Eastern Colorado Health Care System, Denver, Colorado
  - VA Connecticut Healthcare System, New Haven, Connecticut
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - Atlanta VA Health Care System, Atlanta, Georgia
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Nashville VA Medical Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No